CLINICAL TRIAL: NCT02931305
Title: Randomized, Double-blind, Placebo-controlled, Phase 1A Clinical Trial to Assess the Safety, Pharmacokinetic and Pharmacodynamic Effects of Single Escalating Doses of a Standardized Epimedium Prenylflavonoids (EP) Extract (HSA Chinese Proprietary Medicine No: 123317) in Healthy Men.
Brief Title: Epimedium Prenylflavonoid (EP) Extract for Osteoporosis and Cardiovascular Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Obstetrics & Gynaecology, Professor, National University Hospital, Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EP2016
Record Dates: First submitted 2016-10-06; First posted 2016-10-13 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Osteoporosis; Cardiovascular Disease
Keywords: Epimedium prenylflavonoids; Osteoporosis; Cardiovascular diseases; Phase 1; safety; tolerability
MeSH Terms: conditions — Osteoporosis; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epimedium Prenylflavonoids Extract (Experimental): Single oral doses of EP (370 mg, 740 mg and 1110 mg) capsules would be orally administered.
  Interventions: Drug: Epimedium Prenylflavonoids Extract
- Placebo (Placebo Comparator): Single oral doses of Placebo (370 mg, 740 mg and 1110 mg) capsules would be orally administered.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Epimedium Prenylflavonoids Extract — Each Epimedium Prenylflavonoids Extract capsule contains 370 mg of EPIMEDIUM EXTRACT
  Other Names: EP
  Arms: Epimedium Prenylflavonoids Extract
Drug: Placebo — Use iron oxide (brown, black and yellow) to mimic Epimedium Prenylflavonoids Extract.
  Arms: Placebo

SUMMARY:
The primary objective of the trial is to develop Epimedium Prenylflavonoid (EP) extract as a pharmaceutical-quality intervention for post-menopausal osteoporosis and cardiovascular disease. There will be 3 cohorts of 10 healthy men each for the Phase 1 study. In each cohort, 8 men will receive the Epimedium capsules and 2 men will received the matched controls.

DETAILED DESCRIPTION:
Prenylflavonoids and its glycoside derivatives isolated from the Traditional Chinese Medicine (TCM), Epimedium, have potent estrogenic properties. The principal bioactive compounds in Epimedium are the prenylflavonoids, icaritin, and their glycosylated derivatives which can enhance osteoblastic differentiation and mineralization, inhibits bone resorption, and induces apoptosis of osteoclasts. Animal experiments indicate that icariin can prevent bone loss induced by ovariectomized (OVX) in rats, through its stimulatory effects on osteoblast growth and function, and inhibitory action on osteoclast cells.

Epimedium has also demonstrated significant cardiovascular benefits with positive actions on vascular reactivity, endothelial function and thrombosis in human subjects. Notably, icariin, demonstrated a significant nitric oxide (NO)-dependent vasorelaxation of precontracted coronary arterial rings with intact endothelium in a concentration-dependent manner, via the activation of endothelial nitric oxide synthase protein and NO-cyclic guanidine monophosphate (cGMP) pathway. Epimedium prenylflavonoids (EP) can prevent steroid-associated osteonecrosis in rabbit model and notably, reduce thrombosis incidence and shrink fat-cell-size significantly. This striking combination of properties highlights the immense potential in EP for osteoporosis and cardiovascular health.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men.

Exclusion Criteria:

* Hepatitis B patients

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-01 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events/serious adverse events | 8 to10 days
  Incidence and severity of adverse events/serious adverse events based on history, physical examination and vital signs, hematology and clinical chemistry.

SECONDARY OUTCOMES:
lcariin | 3 months
  Serum will be extracted from blood samples for measurement of levels of icariin using Liquid chromatography-mass spectrometry (LC/MS).
Ex vivo osteoblast and osteoclast activities | 6 to 9 months
  Ex vivo assays using human serum to test the effects of EP in bone models of osteoblasts and osteoclasts
Estrogenic biomarkers | 1 to 2 months
  The serum will be tested for cell based estrogen receptor bioassays, and its effects on Michigan Cancer Foundation-7 (MCF-7) cell proliferation will also be assessed.
interleukin-6 (IL-6) | 1 month
  IL-6 assays for thrombosis
high-sensitivity C-reactive protein (hs-CRP) | 1 month
  hs-CRP assays for thrombosis
F2-isoprostanes | 1 month
  F2-isoprostanes assays for thrombosis
multiple platelet aggregation | 1 month
  multiple platelet aggregation assays for thrombosis
Icaritin (ICT) | 3 months
  Serum will be extracted from blood samples for measurement of levels of ICT using LC/MS.
Demethylicaritin (DICT) | 3 months
  Serum will be extracted from blood samples for measurement of levels of DICT using LC/MS.
icariside 1 | 3 months
  Serum will be extracted from blood samples for measurement of levels of icariside 1 using LC/MS.
icariside II | 3 months
  Serum will be extracted from blood samples for measurement of levels of icariside II using LC/MS.

CONTACTS AND LOCATIONS:
Overall Officials: Eu Leong Yong, MD & PhD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- Investigational Medicine Unit, National University Health System, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided